CLINICAL TRIAL: NCT01388777
Title: A Pilot Study to Determine the Efficacy of Cryoablation for the Treatment of Invasive Breast Carcinoma Following Neoadjuvant Therapy
Brief Title: Cryoablation for Invasive Breast Carcinoma Following Neoadjuvant Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination leading to small number of subjects analyzed
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0986; NCI-2011-01278 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Carcinoma; Cryoablation; The Visica 2™ Treatment System; Unifocal primary invasive ductal breast carcinoma; Cryoprobe
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: To determine the rate of complete tumor ablation in patients treated with cryoablation, with complete tumor ablation defined as no remaining invasive or in situ carcinoma present upon pathological examination of the targeted lesion.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Experimental): Cryoablation therapy followed by re-imaging then complete surgical resection.
  Interventions: Device: Visica 2™ Treatment System; Procedure: Cryoablation; Procedure: Surgical Resection

INTERVENTIONS:
Device: Visica 2™ Treatment System — The Visica 2™ Treatment System uses a closed system to circulate liquid nitrogen within the probe tip creating sub-freezing temperatures that result in precision cryoablation of the intended target tissue.
Procedure: Cryoablation — Cryoablation procedure uses a hollow, thin tube called a cryoprobe to freeze and destroy cancer tissue. The cryoprobe needle insertion is done using ultrasound guide to reach target, procedure lasts about 20 minutes.
Procedure: Surgical Resection — Complete surgical resection of the primary tumor following cryoablation therapy.
  Other Names: Surgery

SUMMARY:
Cryoablation is a procedure that uses a hollow, thin tube called a cryoprobe to freeze and destroy cancer tissue.

The goal of this clinical research study is to learn about the level of effectiveness of using ultrasound-guided cryoablation in patients with invasive breast cancer. The safety of this procedure will also be studied.

DETAILED DESCRIPTION:
Study Procedure:

To perform cryoablation in this study, the doctor will insert the cryoprobe like a needle until the tip rests in about the middle of the cancerous area. In this study, an ultrasound imaging device will also be used to allow the doctor to see where to insert the cryoprobe.

If you are found to be eligible and agree to take part in this study, you will have an ultrasound-guided biopsy to confirm your diagnosis. To perform an ultrasound-guided biopsy, a tissue sample will be withdrawn from your breast using a needle and a syringe. A very small amount of tissue will be taken. The needle is guided while being viewed by the doctor on an ultrasound.

Cryoablation:

Before you have the cryoablation procedure, blood (about 1 teaspoon) will be drawn for routine tests. Within 30 days after you join this study, the cryoablation procedure will be performed. The affected area will first be numbed with anesthetic. Your study doctor will insert the cryoprobe needle and use an ultrasound device to help guide the cryoprobe until it reaches the cancerous area.

When in place, the cryoprobe will be used to freeze the cancerous area. The doctor will be very careful to try to avoid damaging the surrounding normal tissue.

The cryoablation procedure will last about 20 minutes. The cryoprobe will be removed when your doctor thinks the cancerous area has been treated as much as possible.

There will be a small wound, like a puncture wound from a large needle. Most likely, you will not need any stitches to close this wound.

First Follow-Up Visit:

About 2-4 weeks after cryoablation:

* You will have a physical exam.
* You will have an MRI scan of the breast to check the status of the disease. This scan is for research purposes only. Researchers want to learn if an MRI scan after cryoablation can detect any remaining breast cancer.

Your MRI scans and the ultrasound images will be reviewed by the study radiologist. This will include the MRI scans from before and after cryoablation, and the ultrasound images from during cryoablation.

Surgery:

Within 4 weeks after cryoablation, you will have standard-of-care surgery to remove the remaining area that was treated during cryoablation. You will be asked to sign a separate consent form that describes the surgery in more detail.

After surgery, the doctor will also check to see if the cryoablation destroyed all of the cancerous area. This will help researchers learn if cryoablation is effective.

Second Follow-Up Visit:

About 2 weeks after surgery:

* You will have a physical exam.
* You will be asked about any side effects you may have had from the cryoablation and surgery.

When you have finished cryoablation and surgery, you and your doctor will decide if you need additional treatment. Additional treatment is not considered part of this study. Your doctor will be able to answer questions you may have about additional treatment.

Length of Study Participation:

You will remain on study for about 2 months. You will be taken off study early if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. The ultrasound-guided cryoablation system that will be used for your cryoablation procedure has been FDA-approved for use in cancer. The use of this system for breast cancer after chemotherapy is investigational.

Up to 10 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Unifocal primary invasive ductal breast carcinoma diagnosed by core needle biopsy. NOTE: Patients with lobular carcinoma, multifocal and/or multicentric ipsilateral breast cancer, multifocal calcifications, or ductal carcinoma in situ (DCIS) with microinvasion are NOT eligible. Patients with contralateral disease will remain eligible.
2. Neoadjuvant chemotherapy or hormonal therapy for the index tumor is required.
3. Residual tumor size </= 2.0 cm in greatest diameter. Specifically, the tumor must measure </= 2.0 cm in the axis parallel to the treatment probe and </= 1.5 cm in the axis anti-parallel to the treatment probe. Largest size measured by mammogram, ultrasound or MRI will be used to determine eligibility.
4. Tumor enhancement on pre-registration MRI.
5. Tumor with <25% intraductal components in the aggregate.
6. Adequate breast size for safe cryoablation. Male breast cancer patients and female breast cancer patients with breasts too small to allow safe cryoablation are not eligible as the minimal thickness of the breast tissue does not lend itself to cryoablation.
7. Patients with prior in-situ or invasive breast carcinomas are eligible if the prior carcinomas occurred in the contralateral breast. Patients with prior in-situ or invasive carcinomas of the ipsilateral breast are not eligible.

Exclusion Criteria:

1. History of open surgical biopsy and/or lumpectomy for diagnosis/treatment of the index breast cancer. Note: Prior rotational and/or vacuum-assisted core biopsies are permitted if no significant distortion is seen on imaging that could obscure visualization and detection of residual disease on MRI, or visualization of cancer on ultrasound for cryoablation procedure.
2. Pregnant and/or lactating. Patients of childbearing potential must have a negative serum or urine pregnancy test. NOTE: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential.
3. Patient has contra-indication to an MRI examination, such as clips/prostheses/implants that are not MRI compatible, or compromised renal function, with a measured or calculated glomerular filtration rate of 60ml/min/1.73m^2
4. Patients less than 18 years of age will not be included in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Hwang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten participants are required for analysis. Patients over 18, with invasive ductal carcinoma with less than or equal to 2 cm residual disease after neoadjuvant treatment, among other criteria are eligible.
Pre-assignment Details: Early termination leading to small number of subjects analyzed.
Groups:
- All Participants Enrolled and Started Treatment: All participants will undergo imaging, cryoablation and further imaging, then surgery.
Period: Overall Study
Arm/Group | All Participants Enrolled and Started Treatment
Started | 1
Cryoablation | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants does not differ from the number of participants assigned to the arms/overall.
Arm/Group | All Participants Enrolled and Started Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Tumor Ablation
Description: The rate of complete tumor ablation in the target lesion will be evaluated by pathologic review of the surgical specimen.
Time Frame: From cryoablation through 30 days from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Enrolled and Started Treatment
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: From cryoablation through 30 days from surgery
Arm/Group | All Participants Enrolled and Started Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT01388777/Prot_SAP_000.pdf